CLINICAL TRIAL: NCT04148664
Title: SHORT-AF: A Randomized Trial of High Power-Short Duration Versus Standard Power-Long Duration Radiofrequency Ablation for Treatment of Atrial Fibrillation
Brief Title: A Trial of High Power-Short Duration Versus Standard Power-Long Duration Radiofrequency Ablation for Treatment of Atrial Fibrillation
Acronym: Short-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHORT-AF
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation Paroxysmal; Atrial Fibrillation, Persistent
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: This is a multi-center prospective single-blinded randomized controlled trial. Enrollment of 60 subjects undergoing clinically-indicated AF ablation is planned with 1:1 block randomization (standard 'low power' RF settings n=30, HPSD n=30 and allowing for 10 drop-outs / consent withdrawals). Follow-up will be over 12 months.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Catheter Settings (Active Comparator): Group 1 - Standard RF ablation settings
  Interventions: Procedure: Catheter ablation with Standard RF ablation settings
- High Power Short Duration (HPSD) (Experimental): Group 2 - High power short duration RF
  Interventions: Procedure: Catheter ablation with High Power Short Duration RF ablation settings

INTERVENTIONS:
Procedure: Catheter ablation with Standard RF ablation settings — Standard RF ablation settings (n=30):
  Maximum 35W for 20-40 seconds, per operator standard.
  Arms: Standard Catheter Settings
Procedure: Catheter ablation with High Power Short Duration RF ablation settings — High power short duration RF (n=30):
  Maximum 50 Watts for 5-15 seconds, per operator standard.
  Arms: High Power Short Duration (HPSD)

SUMMARY:
This study is a prospective, randomized controlled study to compare overall clinical outcomes between High Power Short Duration (HPSD) and standard radiofrequency (RF) ablation settings for Atrial Fibrillation (AF) ablation in the treatment of subjects with paroxysmal or persistent Atrial Fibrillation.

DETAILED DESCRIPTION:
Pulmonary vein isolation using radiofrequency (RF) ablation is a widely used treatment strategy for atrial fibrillation. Peri-procedural complications rates are estimated at between 1.5 - 6% with the two most feared complications being stroke and atrial-esophageal fistula. The risk of these complications increases with (1) longer left atrial dwell times with greater potential for clot formation and (2) esophageal heating during delivery of radiofrequency energy. 'High-power short-duration' (HPSD) is an increasingly utilized strategy to decrease procedure duration and minimize the risk of these complications. Potential mechanisms for benefit include: (1) shorter left atrial dwell times due to more efficient lesion delivery (2) rapid, but more controlled, resistive tissue heating, which avoids deeper, passive conductive heating that can reach the esophagus and cause injury. Moreover, HPSD may improve lesion efficacy and durability due to less recover of excitability after ablation. Despite being widely used and several retrospective studies, there have been no prospective randomized trials comparing outcomes between HPSD and standard RF ablation settings. Moreover, the investigators are interested to see if a shorter procedure (less time in the left atrium) is associated with a lower rate of silent cerebral infarctions (which are occasionally seen on MRI brain post RF ablation - their clinical significance is unclear).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age at their pre-operative visit.
2. Patient is scheduled to have their first AF ablation
3. Paroxysmal or persistent AF
4. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Prior AF ablation
2. Stroke or transient ischemic attack (TIA) within the previous 6 months
3. Known esophageal ulcer or gastrointestinal (GI) bleed within prior 6 months
4. Intent to perform adjunctive left atrial ablation, including posterior wall isolation, left atrial appendage isolation, mitral or other linear lesions.
5. Prior rheumatic heart disease or significant mitral stenosis
6. Mechanical mitral valve replacement
7. Long lasting persistent AF > 1 year
8. Severe left ventricular systolic dysfunction, with LV ejection fraction LVEF<35%
9. Prior left atrial appendage (LAA) occlusion device
10. Prior septal occlusion device
11. Pregnancy
12. Pacemaker, defibrillator or any contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Ablation Duration | During Ablation
  RF ablation duration from start of first pulmonary vein isolation lesion to end of last lesion

SECONDARY OUTCOMES:
Maximum esophageal temperature | During ablation
Maximum esophageal temperature rise | During ablation
Freedom from Atrial Fibrillation | assessed at 6 and 12 months post-ablation
  >30 secs using Ziopatch, 1 year off or on previously ineffective antiarrhythmic drugs (AADs)
Freedom from Atrial Fibrillation | assessed at 6 and 12 months post-ablation
  >30 secs using Ziopatch, 1 year off previously ineffective antiarrhythmic drugs (AADs)
% pulmonary vein pairs isolated with first encirclement | During Ablation
Number of radiofrequency lesions required for isolation/PV | During Ablation
Total left atrial radiofrequency (RF) time | During Ablation
Total procedure duration | During Ablation
Overall complication rate | During Ablation and up to 12 month follow up assessment
Pleurisy | At 1 week and 1 month assessment
Pericardial effusion>1cm | During ablation or up to 30 days post ablation
Pericardial tamponade requiring drainage | During ablation or up to 30 days post ablation
Total saline infused | During Ablation
Presence of asymptomatic cerebral emboli | 1 day post-ablation

CONTACTS AND LOCATIONS:
Overall Officials: Edward P Gerstenfeld, MD, Principal Investigator — Chief of Cardiac Electrophysiology
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
We are open to collaboration but do not plan to give our data to others.

REFERENCES:
- [Background] Perino AC, Leef GC, Cluckey A, Yunus FN, Askari M, Heidenreich PA, Narayan SM, Wang PJ, Turakhia MP. Secular trends in success rate of catheter ablation for atrial fibrillation: The SMASH-AF cohort. Am Heart J. 2019 Feb;208:110-119. doi: 10.1016/j.ahj.2018.10.006. Epub 2018 Oct 29. PMID 30502925
- [Background] Kim TH, Park J, Uhm JS, Joung B, Lee MH, Pak HN. Pulmonary vein reconnection predicts good clinical outcome after second catheter ablation for atrial fibrillation. Europace. 2017 Jun 1;19(6):961-967. doi: 10.1093/europace/euw128. PMID 27256420
- [Background] Asbach S, Biermann J, Bode C, Faber TS. Early Heparin Administration Reduces Risk for Left Atrial Thrombus Formation during Atrial Fibrillation Ablation Procedures. Cardiol Res Pract. 2011;2011:615087. doi: 10.4061/2011/615087. Epub 2011 Jul 2. PMID 21747989
- [Background] Winkle RA, Mohanty S, Patrawala RA, Mead RH, Kong MH, Engel G, Salcedo J, Trivedi CG, Gianni C, Jais P, Natale A, Day JD. Low complication rates using high power (45-50 W) for short duration for atrial fibrillation ablations. Heart Rhythm. 2019 Feb;16(2):165-169. doi: 10.1016/j.hrthm.2018.11.031. PMID 30712645
- [Background] Leshem E, Zilberman I, Tschabrunn CM, Barkagan M, Contreras-Valdes FM, Govari A, Anter E. High-Power and Short-Duration Ablation for Pulmonary Vein Isolation: Biophysical Characterization. JACC Clin Electrophysiol. 2018 Apr;4(4):467-479. doi: 10.1016/j.jacep.2017.11.018. Epub 2018 Feb 2. PMID 30067486
- [Background] Nair KK, Shurrab M, Skanes A, Danon A, Birnie D, Morillo C, Chauhan V, Mangat I, Ayala-Paredes F, Champagne J, Nault I, Tang A, Verma A, Lashevsky I, Singh SM, Crystal E. The prevalence and risk factors for atrioesophageal fistula after percutaneous radiofrequency catheter ablation for atrial fibrillation: the Canadian experience. J Interv Card Electrophysiol. 2014 Mar;39(2):139-44. doi: 10.1007/s10840-013-9853-z. Epub 2013 Dec 7. PMID 24317916
- [Background] Nair KK, Danon A, Valaparambil A, Koruth JS, Singh SM. Atrioesophageal Fistula: A Review. J Atr Fibrillation. 2015 Oct 31;8(3):1331. doi: 10.4022/jafib.1331. eCollection 2015 Oct-Nov. PMID 27957213
- [Background] Han HC, Ha FJ, Sanders P, Spencer R, Teh AW, O'Donnell D, Farouque O, Lim HS. Atrioesophageal Fistula: Clinical Presentation, Procedural Characteristics, Diagnostic Investigations, and Treatment Outcomes. Circ Arrhythm Electrophysiol. 2017 Nov;10(11):e005579. doi: 10.1161/CIRCEP.117.005579. PMID 29109075
- [Background] Bhaskaran A, Chik W, Pouliopoulos J, Nalliah C, Qian P, Barry T, Nadri F, Samanta R, Tran Y, Thomas S, Kovoor P, Thiagalingam A. Five seconds of 50-60 W radio frequency atrial ablations were transmural and safe: an in vitro mechanistic assessment and force-controlled in vivo validation. Europace. 2017 May 1;19(5):874-880. doi: 10.1093/europace/euw077. PMID 27207815
- [Background] Baher A, Kheirkhahan M, Rechenmacher SJ, Marashly Q, Kholmovski EG, Siebermair J, Acharya M, Aljuaid M, Morris AK, Kaur G, Han FT, Wilson BD, Steinberg BA, Marrouche NF, Chelu MG. High-Power Radiofrequency Catheter Ablation of Atrial Fibrillation: Using Late Gadolinium Enhancement Magnetic Resonance Imaging as a Novel Index of Esophageal Injury. JACC Clin Electrophysiol. 2018 Dec;4(12):1583-1594. doi: 10.1016/j.jacep.2018.07.017. Epub 2018 Sep 26. PMID 30573123